CLINICAL TRIAL: NCT05802095
Title: The Effect of Supplemental Feeding Tube Devices Used in Preterms on Baby's Breastfeeding Success and Mother's Breastfeeding Self-Efficacy
Brief Title: Effect of Supplemental Feeding Tube Devices in Breastfeeding Success and Mother's Breastfeeding Self-Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Hilal Berber Çiftci, İstanbul Medipol University, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Urfa
Record Dates: First submitted 2023-03-24; First posted 2023-04-06 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Breastfeeding; Feeding Disorder Neonatal
Keywords: neonatal feeding; breastfeeding; supplemental feeding tube device
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Clinical Trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The babies in the experimental group are fed 3 meals from the day after the decision to switch to oral feeding, with supplemental feeding tube device(SFTD) (09:00-12:00-15:00) and other meals with a bottle.
  Interventions: Device: Supplemental Feeding Tube Device
- Control (No Intervention): The babies in the control group, on the other hand, will be fed 3 meals a day (09:00-12:00-15:00) after the decision to switch to oral feeding, which is the routine feeding method of the intensive care unit, and with a bottle for other meals in the same way.

INTERVENTIONS:
Device: Supplemental Feeding Tube Device — One end of the catheter is in such a way that milk comes into the bottle. The tip of the feeding catheter can be fixed to the mother's breast with a plaster so that it is in the baby's mouth. The tip of the catheter is placed inside the baby's mouth while the baby is sucking on its mother. While the mother is breastfeeding, milk is supplied to the baby from both the mother and the bottle. The baby will continue to suckle as he feels that plenty of milk is coming. To increase the flow of milk from the bottle, the mother hangs the bottle around her neck with the teat side down. The higher the bottle or milk container is held, the greater the flow of milk. It is an easy and safe method.
  Arms: Experimental group

SUMMARY:
The research will be carried out as a randomized controlled experimental design to evaluate the effectiveness of the breastfeeding support system to increase sucking success in premature infants receiving care in the NICU and breastfeeding self-efficacy in mothers.

In the study, the experimental and control groups will be determined by randomization of premature babies hospitalized in the NICU. While the babies in the control group will be fed with the routine feeding method (bottle) of the NICU, the babies in the experimental group will be fed with the breastfeeding support system by their mother. Research data will be collected using the Premature Baby and Its Mother Information Form, Premature Baby Follow-up Form, LATCH Breastfeeding Diagnostic Scale and Breastfeeding Self-Efficacy Scale-Short Form.

DETAILED DESCRIPTION:
Premature babies have to cope with many problems in the neonatal intensive care unit (NICU) in the postnatal period, and feeding problems are the leading of these problems. Oral feeding of premature infants is a complex and dynamic process consisting of the interaction of oral-motor, neurological, cardiorespiratory and gastrointestinal systems. Because they are anatomically and physiologically immature, they often cannot coordinate their sucking, swallowing and respiration for oral feeding, and they often have difficulty in oral feeding. Therefore, feeding premature babies in the NICU is provided by an orogastric or nasogastric tube. Continuing the feeding with the gavage method for a long time causes a delay in the acquisition of the motor skills required for oral feeding. Therefore, premature babies should be switched to oral feeding when they are physiologically ready. It is known that growth and developmental retardation are seen in premature babies if appropriate and adequate nutrition is not provided on time.

The most basic criterion sought in the transition to oral feeding in premature babies is the development of feeding skills. Different oral stimulus interventions have been developed to support and strengthen the development of oral-motor functions, create sufficient suction power, and start oral nutrition earlier. Tactile/kinesthetic stimulation, oral stimulation, swallowing exercises, non-nutritive sucking, gentle pressure on the cheeks, lips, chin and palate are among the most common sensorimotor interventions. It is reported that these interventions accelerate the transition time to oral feeding. Successful sucking transition from gavage to full oral feeding is one of the most important determinants of both discharges from the NICU and the growth and development of premature infants. This study will evaluate the effect of the breastfeeding support system used in premature babies on the baby's sucking success and the mother's breastfeeding self-efficacy.

The research will be carried out as a randomized controlled experimental design to evaluate the effectiveness of the breastfeeding support system to increase sucking success in premature infants receiving care in the NICU and breastfeeding self-efficacy in mothers.

In the study, the experimental and control groups will be determined by randomization of premature babies hospitalized in the NICU. While the babies in the control group will be fed with the routine feeding method (bottle) of the NICU, the babies in the experimental group will be fed with the breastfeeding support system by their mother. Research data will be collected using the Premature Baby and Its Mother Information Form, Premature Baby Follow-up Form, LATCH Breastfeeding Diagnostic Scale and Breastfeeding Self-Efficacy Scale-Short Form.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenstrual age 32 and 35 weeks of gestation,
2. Over 1500 g,
3. Switching to oral feeding after feeding with orogastric tube,
4. Who has been breastfed during gavage feeding,
5. Those who have not completed the first 24 hours in the transition from oragastric tube feeding to the oral feeding process,
6. Having cues of readiness for feeding (tolerating enteral nutrition, having a stable oxygen saturation and breathing during feeding, having the ability to lick, swallow and suck, react when mouth and lip are given stimuli),
7. The mother's willingness to breastfeed her baby,
8. Premature babies of parents who volunteered to participate in the study will be included.

Exclusion Criteria:

1. Having diseases other than being premature
2. Able to successfully take the breast in the first attempt,
3. Congenital anomaly,
4. Chromosomal disorders,
5. Having sepsis
6. With intracranial bleeding,
7. Those with a very low birth weight below 1500 g and
8. Less than 32nd gestational week,
9. Premature babies older than 35 weeks of gestation will be excluded.

Ages: 32 Weeks to 35 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
LATCH a breastfeeding charting system and documentation tool | 1 hours
  LATCH is a diagnostic tool whose scoring system is similar to the Apgar score system. The scale consists of five evaluation criteria. The LATCH diagnostic tool is formed from the English initials of these five criteria. For each criterion that makes up the LATCH Breastfeeding Diagnostic and Evaluation Scale, 0,1, 2 points are given. Breastfeeding success is evaluated by summing the scores. The highest score that can be obtained from the scale is 10 and the lowest score is 0. The higher the score obtained from the scale, the higher the success of breastfeeding. In the research, the mother and her baby will be observed and evaluated while breastfeeding.
Breastfeeding Self-Efficacy Short Form Scale | 1 hours
  The scale is in 5-point Likert type and the items of the scale are evaluated by grading from 1 "I am not sure" to 5 "I am always sure". The lowest score that can be obtained from the scale is 14, and the highest score is 70. A high score on the scale indicates higher breastfeeding self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Bozdağ, Principal Investigator — Harran University
Locations (1):
- Şanlıurfa Eğitim ve Araştırma Hastanesi, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Celik F, Sen S, Karayagiz Muslu G. Effects of Oral Stimulation and Supplemental Nursing System on the Transition Time to Full Breast of Mother and Sucking Success in Preterm Infants: A Randomized Controlled Trial. Clin Nurs Res. 2022 Jun;31(5):891-900. doi: 10.1177/10547738211058312. Epub 2021 Nov 16. PMID 34784787